CLINICAL TRIAL: NCT00223873
Title: The Use of Penile Vibratory Stimulation to Decrease Spasticity Following Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7927-09
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-05

CONDITIONS: Spinal Cord Injury; Muscle Spasticity
Keywords: Penile Vibratory Stimulation; Muscles Spasticity; Spasms; Ferti Care Vibrator; Antispasmotic treatment
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Spasm

INTERVENTIONS:
Procedure: Penile Vibratory Stimulation

SUMMARY:
The purpose of this study is to determine the effect of penile vibratory stimulation on the muscle spasticity of men with chronic spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury can result in mild to severe muscle spasms that can both inhibit functional capability and increase the likelihood of injury due to fall. Anecdotal reports and a recent study suggest that triggering the ejaculatory reflex in men with vibratory stimulation can result in a significant decrease in spasm activity over a period of 2 to 42 hours. This study examines the effects of penile vibratory stimulation on spasticity when conducted daily in the home setting.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with a traumatic spinal cord injury

* Level of injury is at T6 or below
* Injured at least 6 months prior to study enrollment
* Male, aged 18 to 70 years
* Spasticity to a degree that either anti-spasticity medications have been or are being used or current spasticity is at 2 or greater on the Ashworth scale specifically for the quadriceps muscle group (knee flexion)

Exclusion Criteria:

* Medical instability
* Subjects may not use Cialis
* Use of Viagra, Levitra, Caverject, or vacuum constriction devices is restricted to no less than 8 hours prior to daily vibratory therapy
* Recent history of autonomic dysreflexia secondary to sexual stimulation
* Presence of intrathecal Baclofen pumps
* Inability or unwillingness to use the therapy daily

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Spasticity in the lower extremities will be scored per the
Ashworth scale at each weekly visit. Additionally,
subjects will record their daily spasm frequency on a 5
point scale in the form of a daily questionnaire. Intra
and inter-visit indicies of spas.

SECONDARY OUTCOMES:
Several questionnaires such as the CHART, SWLS, FIM, and IIEF are used to assess changes in quality of life and function.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo E Gousse, MD, Principal Investigator — Miami VA Medical Center Urology Service
Locations (1):
- Miami Veterans Affairs Medical Center, Miami, Florida, United States

REFERENCES:
- [Background] Maynard FM, Karunas RS, Waring WP 3rd. Epidemiology of spasticity following traumatic spinal cord injury. Arch Phys Med Rehabil. 1990 Jul;71(8):566-9. PMID 2369291
- [Background] Zierski J, Muller H, Dralle D, Wurdinger T. Implanted pump systems for treatment of spasticity. Acta Neurochir Suppl (Wien). 1988;43:94-9. doi: 10.1007/978-3-7091-8978-8_21. PMID 3213666
- [Background] Young RR, Delwaide PJ. Drug therapy: spasticity (first of two parts). N Engl J Med. 1981 Jan 1;304(1):28-33. doi: 10.1056/NEJM198101013040107. No abstract available. PMID 6448959
- [Background] Penn RD, Savoy SM, Corcos D, Latash M, Gottlieb G, Parke B, Kroin JS. Intrathecal baclofen for severe spinal spasticity. N Engl J Med. 1989 Jun 8;320(23):1517-21. doi: 10.1056/NEJM198906083202303. PMID 2657424
- [Background] Knutsson E, Lindblom U, Martensson A. Plasma and cerebrospinal fluid levels of baclofen (Lioresal) at optimal therapeutic responses in spastic paresis. J Neurol Sci. 1974 Nov;23(3):473-84. doi: 10.1016/0022-510x(74)90163-4. No abstract available. PMID 4154365
- [Background] Ochs G, Struppler A, Meyerson BA, Linderoth B, Gybels J, Gardner BP, Teddy P, Jamous A, Weinmann P. Intrathecal baclofen for long-term treatment of spasticity: a multi-centre study. J Neurol Neurosurg Psychiatry. 1989 Aug;52(8):933-9. doi: 10.1136/jnnp.52.8.933. PMID 2487035